CLINICAL TRIAL: NCT04032249
Title: Implications of Self-weighing During Weight Loss Treatment: A Pragmatic 6-month Randomized Trial
Brief Title: Implications of Self-weighing During Weight Loss Treatment
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Alberto Hernández de los Reyes, Principal Investigator, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: P5_A284R4156
Record Dates: First submitted 2019-07-22; First posted 2019-07-25 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2019-07

CONDITIONS: Overweight and Obesity; Signs and Symptoms; Behavior, Eating
Keywords: Obesity; Self-weighing; Weight loss; Mobile health
MeSH Terms: conditions — Overweight; Obesity; Signs and Symptoms; Feeding Behavior; Weight Loss | interventions — Control Groups

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (CG) (Active Comparator): Education and modifying diet
  Interventions: Behavioral: Control Group (CG)
- Intervention Group (IG) (Experimental): Education, modifying diet and Indications to record self-weighing with a frequency of 2 times per week
  Interventions: Behavioral: Intervention Group (IG)

INTERVENTIONS:
Behavioral: Control Group (CG) — The control group is subjected to follow a hypocaloric diet and receives information about the benefits of having healthy habits in relation to decision making and food
  Arms: Control Group (CG)
Behavioral: Intervention Group (IG) — The control group is subjected to follow a hypocaloric diet and receives information about the benefits of having healthy habits in relation to decision making and food, but also, they will have monitored the self-control of the weight in order to compare the impact of self-weighing versus not doing it
  Arms: Intervention Group (IG)

SUMMARY:
This study aims to analyze the effectiveness of introducing behavioral elements in a weight loss program, in this case, comparing the difference between self-weighing versus not doing so.

ELIGIBILITY:
Inclusion Criteria:

* Having a IMC >25,
* Being sedentary and
* Have not been submitted to a restrictive diet in the 6 months preceding this study

Exclusion Criteria:

* Suffered from type 2 diabetes or renal conditions
* Being pregnancy or attempt at pregnancy,
* Undergoing antidepressant pharmacological treatment

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — the present study is carried out in men
Enrollment: 70 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-12-15 (Actual); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline BMI | At baseline (0 years) and followed for 2 years
  Baseline mean BMI values will be measured and compared at 3, 6, 12 and 24 months. BMI will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale
Changes from baseline Fatty mass | At baseline (0 years) and followed for 2 years
  Baseline mean Fatty mass values will be measured and compared at 3, 6, 12 and 24 months. Fatty mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a percentage.
Changes from baseline Free-fatty mass | At baseline (0 years) and followed for 2 years
  Baseline mean Free-fatty mass values will be measured and compared at 3, 6, 12 and 24 months. Free-fatty mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a percentage.
Changes from baseline Muscular Mass | At baseline (0 years) and followed for 2 years
  Baseline mean Muscular Mass values will be measured and compared at 3, 6, 12 and 24 months. Muscular Mass will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a Kg.
Changes from baseline Corporal Water | At baseline (0 years) and followed for 2 years
  Baseline mean Corporal Water values will be measured and compared at 3, 6, 12 and 24 months. Corporal Water will be assessed on a monthly basis during nutritional consultation through a Bioelectrical Impedance Analysis method using a Tanita BC-418 Segmental Body Composition Analyser/Scale. Fatty mass is measured as a Kg.
Adherence to dietary pattern will be also measured through personal interview | At baseline (0 years) and followed for 2 years
  Participants will be subjected for an intervention based on nutritional (control group) and physical education (two intervention arms) during 24 months. Partial measures will be also taken every week. In the end of the trial, changes in dietary patterns will be measured comparing means differences between baselines, 3, 6, 12 and 24 months.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad de Córdoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hernandez-Reyes A, Camara-Martos F, Vidal A, Molina-Luque R, Moreno-Rojas R. Effects of Self-Weighing During Weight Loss Treatment: A 6-Month Randomized Controlled Trial. Front Psychol. 2020 Mar 10;11:397. doi: 10.3389/fpsyg.2020.00397. eCollection 2020. PMID 32210897